CLINICAL TRIAL: NCT07128303
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GS-5319 in Adults With MTAP-deleted Advanced Solid Tumors
Brief Title: Study of GS-5319 in Adults With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-707-7297
Record Dates: First submitted 2025-08-13; First posted 2025-08-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: GS-5319 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of GS-5319 monotherapy, until disease progression, or until the participants meets other study drug discontinuation criteria as specified in protocol or up to 105 weeks, whichever occurs first to determine the recommended dose for dose expansion phase.
  Interventions: Drug: GS-5319
- Part B: GS-5319 Monotherapy Dose Expansion (Experimental): Participants will be enrolled in different cohorts based on the selected indications to receive GS-5319 monotherapy at the recommended dose during the monotherapy dose expansion phase.
  Interventions: Drug: GS-5319

INTERVENTIONS:
Drug: GS-5319 — Administered orally

SUMMARY:
The goal of this clinical study is to learn more about the study drug, GS-5319, its dosing, safety and tolerability in adults with solid tumors, where the participants show a specific gene alteration in the tumor. The gene helps produce methylthioadenosine phosphorylase (MTAP) enzyme. MTAP enzyme helps in normal growth of cells.

The primary objectives of the study are to assess the safety and tolerability of GS-5319 in participants with methylthioadenosine phosphorylase (MTAP)-deleted advanced solid tumors and to identify the maximum tolerated dose (MTD)/maximum administered dose (MAD) and/or the recommended dose for expansion (RDE).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants diagnosed with histologically or cytologically confirmed solid tumor types who have progressed despite standard therapy, are intolerant to standard therapy, or are ineligible for standard therapy in the advanced setting (locally-advanced or metastatic).
* Participant tumors are methylthioadenosine phosphorylase (MTAP)-deficient. Deoxyribonucleic acid (DNA) sequencing may be assessed locally such as by local next-generation sequencing (NGS) or by central laboratory assay when available.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* Adequate organ function
* Age ≥ 18yrs old ( ≥ 19 years old for patients in South Korea)
* Participants must meet the following tissue requirements:

  1. Part A and B: pretreatment tumor tissue is required

Key Exclusion Criteria:

* Active second malignancy. Participants with a history of malignancy who have been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or participants with surgically cured tumors with low risk of recurrence may be enrolled.
* Positive serum pregnancy test or participant who is breastfeeding.
* Requirement for ongoing therapy with any prohibited medications.
* Have not recovered (ie, returned to Grade 1 or baseline) from adverse events (AEs) due to a previously administered agent.
* Active and clinically relevant bacterial, fungal, or viral infection that is not controlled or requires systemic antibiotics, antifungals, or antivirals, respectively.
* Ascites or pleural effusion that is symptomatic and/or requiring medical intervention.
* Active human immunodeficiency virus (HIV)/hepatitis B virus (HBV)/hepatitis C virus (HCV) infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serous Adverse Events (SAEs) | First Dose up to 30 days post last dose (Up to 105 weeks)
Percentage of Participants Experiencing Laboratory Abnormalities | First Dose up to 30 days post last dose (Up to 105 weeks)
Percentage of Participants Experiencing any Dose-limiting Toxicities (DLTs) in Dose-escalation Cohorts | Up to 21 days

SECONDARY OUTCOMES:
Plasma Concentration of GS-5319 | Predose and postdose up to end of treatment (up to 105 weeks)
Pharmacokinetic (PK) parameter: AUC0-24 of GS-5319 | Predose and postdose up to end of treatment (up to 105 weeks)
  AUC0-24 is defined as the partial area under the concentration versus time curve from time 0 to time 24 hours.
PK parameter: Cmax of GS-5319 | Predose and postdose up to end of treatment (up to 105 weeks)
  Cmax is defined the maximum observed plasma drug concentration.
PK parameter: Tmax of GS-5319 | Predose and postdose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (7):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - START San Antonio, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid - FJD - Hospital Fundación Jiménez Díaz - Phase I Clinical Trials Unit, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT07128303